CLINICAL TRIAL: NCT05677867
Title: A PHASE 1, OPEN-LABEL, 2-PERIOD, 2-SEQUENCE, CROSSOVER STUDY TO COMPARE THE SINGLE-DOSE PHARMACOKINETICS OF 2 DIFFERENT FORMULATIONS OF PF-07081532 ADMINISTERED ORALLY TO ADULT PARTICIPANTS WHO ARE OVERWEIGHT OR OBESE
Brief Title: A Study to Compare Two Different Forms of PF-07081532 in Adults Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3991010
Record Dates: First submitted 2022-12-13; First posted 2023-01-10 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Overweight; Obesity
Keywords: PF-07081532
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: PF-07081532 80 mg will be provided in 2 different oral formulations (A and B). Formulation A will be administered as a PF-07081532 20 mg immediate release tablet and a 60 mg immediate release tablet. Formulation B will be administered as a PF-07081532 80 mg immediate release tablet. The overall design is a randomized, open-label, single dose, 2-period, 2-sequence, crossover study.
Masking Description: (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Formulation A (Reference) followed by Formulation B (Test) (Experimental)
  Interventions: Drug: Formulation A (PF-07081532 20 mg plus 60 mg); Drug: Formulation B (PF-07081532 80 mg)
- Formulation B (Test) followed by Formulation A (Reference) (Experimental)
  Interventions: Drug: Formulation A (PF-07081532 20 mg plus 60 mg); Drug: Formulation B (PF-07081532 80 mg)

INTERVENTIONS:
Drug: Formulation A (PF-07081532 20 mg plus 60 mg) — Formulation A: administered as a 20 mg immediate release tablet and a 60 mg immediate release tablet
Drug: Formulation B (PF-07081532 80 mg) — Formulation B: administered as a 80 mg immediate release tablet

SUMMARY:
The purpose of this study is to compare the amount of PF-07081532 in blood after taking two different forms of PF-07081532. This study is seeking participants who are at least 18 years of age and are overweight and/or obese. All study participants will receive a total of 2 single doses of this study medication in either form. Form A consists of a PF-07081532 20 mg immediate release tablet and a PF-07081532 60 mg immediate release tablet. Form B consists of a PF-07081532 80 mg immediate release tablet. Each single dose will be separated by a minimum of 6 days. The amount of PF-07081532 in the blood for 4 days after taking each single dose will be compared between the two different formulations of PF-07081532.

The total time that participants will take part in this study is about 70 days. The first visit is a screening visit to ensure that participants are appropriately qualified for the study. This will occur up to 28 days before the first single dose. Participants will be admitted into the clinic one day prior to the first single dose and will remain in the clinic for a total of 11 days. The study team will phone the participants 28 to 35 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be at least 18 years of age, inclusive, at the time of signing the ICD
* Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and ECGs
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
* A total body weight >50 kg (110 lb) and BMI of 25.0 to <34.9 kg/m2, inclusive, at the screening visit
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and protocol

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing)
* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection)
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2, or pancreatitis, or participants with suspected MTC per the investigator's judgement
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention
* In females, current use of hormone replacement therapy or oral/injectable contraceptives containing ethinyl estradiol
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) preceding the first dose of study intervention used in this study. Investigational products which are strong CYP3A inducers or time-dependent inhibitors are prohibited within 14 days plus 5 half-lives or 30 days (whichever is longer) prior to the dose of study intervention
* Known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving PF-07081532 or known intolerance to a GLP-1R agonist
* A positive urine drug test
* Using a properly sized and calibrated BP cuff, screening supine BP ≥140 mm Hg (systolic) or 90 mm Hg (diastolic) following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility
* Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate- age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:
* Aspartate aminotransferase or alanine aminotransferase level ≥1.25 × upper limit of normal (ULN);
* Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN;
* HbA1c ≥6.5%;
* Fasting blood glucose ≥126 mg/dL (7 mmol/L);
* Calcitonin > ULN;
* eGFR <60 mL/min/1.73 m2 as calculated by the CKD-EPI equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were enrolled and treated in the study. All 20 participants completed the study.
Groups:
- Sequence 1: Participants in Sequence 1 received a single dose of PF-07081532 20 mg immediate release tablet and 60 mg immediate release tablet (Formulation A) on Period 1 Day 1, and then received a single dose of PF-07081532 80 mg immediate release tablet (Formulation B) on Period 2 Day 1, with a minimum washout period of 6 days between the 2 doses.
- Sequence 2: Participants in Sequence 2 received a single dose of PF-07081532 80 mg immediate release tablet (Formulation B) on Period 1 Day 1, and then received a single dose of PF-07081532 20 mg immediate release tablet and 60 mg immediate release tablet (Formulation A) on Period 2 Day 1, with a minimum washout period of 6 days between the 2 doses.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This group includes all participants who enrolled in this study and received at least 1 dose of study intervention regardless of the arms they assigned to.
Groups:
- All Participants: This group includes all participants who enrolled in this study and received at least 1 dose of study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.90 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Median (Full Range); unit: kg/m^2] — BMI is a person's weight in kilograms divided by the square of height in meters.
  kg/m^2 | 28.55 [25.4 to 32.6]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Parameter - Area Under the Concentration-Time Curve to Infinity (AUCinf) of PF-07081532
Description: AUCinf is the area under the concentration-time curve to infinity. AUCinf was calculated by AUClast + (Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours post dose on Day 1 of Period 1 and Period 2
Population: All participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here "Number of Participants Analyzed" signifies participants who contributed to this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Formulation A: Formulation A was administrated as PF-07081532 20 mg immediate release tablet and 60 mg immediate release tablet. Participants in Sequence 1 received Formulation A in Period 1, participants in Sequence 2 received Formulation A in Period 2.
- Formulation B: Formulation B was administrated as PF-07081532 80 mg immediate release tablet. Participants in Sequence 1 received Formulation B in Period 2, participants in Sequence 2 received Formulation B in Period 1.
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 17 | 18
nanogram*hour/milliliter (ng*hr/mL) | 179400 (40) | 178300 (49)
Statistical Analysis 1: Comparison: Formulation A vs Formulation B; Natural log transformed AUCinf was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect. The adjusted mean differences and 90% Confidence Intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. Formulation A was the Reference treatment while Formulation B was the Test treatment; Test type: Other; Ratio of Adjusted Geometric Means = 97.40, 90% CI 2-sided [92.92 to 102.08] — The ratios (and 90% CIs) are expressed as percentages

2. Primary Outcome: Pharmacokinetics Parameter - Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07081532
Description: AUClast is the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast was calculated by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Formulation A: Formulation A was administrated as PF-07081532 20 mg immediate release tablet + 60 mg immediate release tablet. Participants in Sequence 1 received Formulation A in Period 1, participants in Sequence 2 received Formulation A in Period 2.
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 17 | 18
ng*hr/mL | 171900 (38) | 170400 (47)
Statistical Analysis 1: Comparison: Formulation A vs Formulation B; Natural log transformed AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. Formulation A was the Reference treatment while Formulation B was the Test treatment; Test type: Other; Ratio of Geometric Adjusted Means = 97.36, 90% CI 2-sided [92.77 to 102.17] — The ratios (and 90% CIs) are expressed as percentages

3. Primary Outcome: Pharmacokinetics Parameter - Maximum Observed Concentration (Cmax) of PF-07081532
Description: Cmax is the maximum observed concentration.
Time Frame: Pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, and 96 hours post dose of Day 1 Period 1 and Period 2.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 17 | 18
nanogram/milliliter (ng/mL) | 8072 (29) | 7741 (27)
Statistical Analysis 1: Comparison: Formulation A vs Formulation B; Natural log transformed Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within the sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. Formulation A was the Reference treatment while Formulation B was the Test treatment; Test type: Other; Ratio of Adjusted Means = 94.70, 90% CI 2-sided [81.40 to 110.18] — The ratios (and 90% CIs) are expressed as percentages

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All-Causality and Treatment-Related)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. Treatment-emergent are events between first dose of study intervention and up to 28-35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose up to 28 to 35 days after administration of the final dose of study intervention (maximum of 51 days)
Population: All participants who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 20 | 20
Participants
  All Causality TEAEs | 9 | 8
  Treatment-Related TEAEs | 9 | 8
  All-Causality Treatment-Emergent SAE | 0 | 0
  Treatment-Related Treatment-Emergent SAE | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants with laboratory abnormalities that met pre-specified criteria: Urate (millimole/Liter) > 1.2*ULN (upper limit of normal) and Monocytes/Leukocytes (%) > 1.2*ULN.
Time Frame: Baseline (Day 1) up to Period 2 Day 5
Population: All participants who took at least 1 dose of study intervention. Here "Number of Participants Analyzed" signifies participants who contributed to this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 10 | 10
Participants
  Monocytes/Leukocytes (%) > 1.2*ULN | 0 | 1
  Urate (mmol/L) > 1.2*ULN | 0 | 1

6. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria of Vital Signs
Description: Pre-specified criteria of vital signs included: Systolic blood pressure (BP): minimum (min) <90 mmHg, change from baseline (CfB) maximum (max) decrease or increase >=30mmHg; Diastolic BP min <50mmHg, CfB max decrease or increase >=20mmHg; supine pulse rate: min < 40 beats per minute (bpm), max > 120 bpm.
Time Frame: Baseline (Day 1) up to Period 2 Day 5
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Meeting Pre-Specified Criteria of Electrocardiogram (ECGs)
Description: The pre-specified criteria of ECG included: PR interval, aggregated: value >=300 msec, %change >= 25/50% msec; QRS duration, aggregated: value>=200 msec, %changes >= 25/50% msec; QTCF interval, aggregated: 450<=value<480 msec, 480<=value<500 msec, value>=500 msec, 30<=changes<60msec, and changes>=60msec.
Time Frame: Baseline (Day 1) up to Period 2 Day 5
Population: All participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A | Formulation B
Number analyzed (Participants) | 20 | 20
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first dose up to 28 to 35 days after administration of the final dose of study intervention (maximum of 51 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Formulation A | Formulation B
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Formulation A (N=20) | Formulation B (N=20)
Constipation (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 7 | 7
Vomiting (Gastrointestinal disorders) | 3 | 3
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT05677867/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT05677867/SAP_001.pdf